CLINICAL TRIAL: NCT02478138
Title: Sentinel Lymph Node Mapping of Oral Cancer Using Near-Infrared Fluorescence Imaging
Acronym: SLN Mapping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-7441
Record Dates: First submitted 2015-06-01; First posted 2015-06-23 (Estimated); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Indocyanine Green; Diagnostic Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surgical - therapeutic (Other): patients will be enrolled under informed consent based upon their medical diagnosis, planned surgical procedures, and suitability for the procedure. During the study, patients will receive injections of ICG and will be imaged using a commercial NIR imaging system
  Interventions: Procedure: Sentinel lymph node mapping; Drug: Indocyanine Green (ICG); Device: near-infrared fluorescence (NIR) imaging (Pinpoint, Novadaq, Waterloo)

INTERVENTIONS:
Procedure: Sentinel lymph node mapping — Thirty (30) patients will be enrolled under informed consent based upon their medical diagnosis, planned surgical procedures, and suitability for the procedure. During the study, patients will receive injections of ICG and will be imaged using a commercial NIR imaging system (Pinpoint, Novadaq, Waterloo ON). After the study, patients will continue with their planned management.
  Other Names: near-infrared (NIR) fluorescent dye indocyanine green
Drug: Indocyanine Green (ICG)
Device: near-infrared fluorescence (NIR) imaging (Pinpoint, Novadaq, Waterloo)

SUMMARY:
Cervical lymph node involvement, in head and cancer neck patients, is one of the most important prognostic factors. Currently patients undergo neck dissection removing some or all nodes and neck involvement is retrospectively determined. Sentinel lymph node (SLN) identification and biopsy has become clinical practise in other areas including breast, skin, and gastric cancer. The gold standard for detecting metastatic lymph nodes is pathological analysis, but the lack of an accurate or clinically accepted way to identify sentinel lymph nodes in the cervical region has motivated the usage of indocyanine green (ICG) and near-infrared fluorescence (NIR) imaging (Pinpoint, Novadaq, Waterloo). A prospective clinical trial using a commercially available NIR system and ICG injection around the tumour site will evaluate the ability to detect and biopsy sentinel lymph nodes in head and neck cancer patients.

DETAILED DESCRIPTION:
Clinical systems for fluorescence imaging using ICG have recently been published with reported SLN identification rates of 94-100% in breast and colorectal cancers. The traditional radioisotope method enables navigation to the site of skin incision by measurement of radiation uptake, whereas the ICG fluorescence method can precisely identify the site of skin incision by tracing the lymphatic vessels across the skin and without radiation exposure. Systematic reviews have shown that the incidence of false negative SLN biopsy is high in head and neck applications. Therefore, the fluorescence SLN method, can potentially provide more precise information regarding which lymph nodes should be removed. As the ICG fluorescence technique can identify the basin that includes not only SLNs but also para-SLNs where the lymphatic vessels drain, the average number of lymph nodes removed also tends to increase. In preliminary studies, the ICG technique achieves a high identification rate comparable to that of the radioactive method. There has been to date, however, only limited studies of this technique in the area of oral cancer lymph node mapping. In our study we propose to evaluate the potential application of ICG in the mapping and detection of SLN in cancers of the head and neck in comparison with the radioactive agent method. We hypothesize that NIR-guided SLNB could present a new, safe and sensitive alternative or addition to the conventional SLN procedure.

ELIGIBILITY:
Inclusion Criteria:

* The study will include patients with tumors or other masses in the following sites: oral cavity, oropharynx, nasal cavity, sinuses, nasopharynx, parapharyngeal space, parotid salivary glands, head and neck skin and skull base.
* N0 neck status
* The patients should have a complete and detailed medical record.
* Subjects must be at least 18 years of age.
* Subjects must sign and be given a copy of the written Informed Consent Form.

Exclusion Criteria:

* Patients who are not able to consent by themselves or grasp the implication of the study.
* Subjects participating in any other clinical trial during the time of this clinical investigation and that may have an impact on this evaluation.
* Pregnant or potentially pregnant woman
* Lactation.
* Iodine, shellfish, cough mixture, betadine or ICG allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-05; Primary Completion 2024-01-08 (Actual); Study Completion 2024-01-08 (Actual)

PRIMARY OUTCOMES:
ICG imaging to identify lymph nodes metastases in head and neck cancer | During surgical procedure
  The aim of this proposal is to evaluate the potential application of Indocyanine Green (ICG) in the mapping and detection of sentinel lymph nodes (SLN) in cancers of the head and neck.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan C Irish, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada